CLINICAL TRIAL: NCT01181752
Title: Educational Intervention, Observing Participants' Proficiency of Eye Drop Instillation
Brief Title: Proficiency of Eye Drop Instillation in Postoperative Cataract Patients in Ghana
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-01479
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Cataract Surgery
Keywords: proficiency; eye drop instillation; postoperative cataract surgery; Ghana

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group A: Baseline/control subjects who are only tested on postoperative day 30
- Group B: Subjects who will be tested on postoperative day 1 and day 30
- Group C: Subjects who cannot proficiently administer the medication on postoperative day 1 will be re-classified as "Group C" subjects

SUMMARY:
Eye drops must be proficiently instilled to prevent infections following cataract surgery. Proficiency is defined as placing a drop on the ocular surface without touching the applicator's tip. Researchers will investigate whether patients can proficiently administer eye drops on the first attempt on the first day after surgeries. If successful, researchers will determine how proficient they are 29 days later. If not, they will be provided with additional educational sessions and tested again 29 days later. Researchers will also determine if the proficiency of instillation correlates to whether patients experience irritation or pain after surgery.

Summary Brief Summary Eye drops must be proficiently instilled to prevent infections following cataract surgery. Proficiency is defined as placing a drop on the ocular surface without touching the applicator's tip. Researchers will investigate whether patients can proficiently administer eye drops on the first attempt on the first day after surgeries. If successful, researchers will determine how proficient they are 29 days later. If not, they will be provided with additional educational sessions and tested again 29 days later. Researchers will also determine if the proficiency of instillation correlates to whether patients experience irritation or pain after surgery.

Hypotheses:

On postoperative day 30, there will be a higher rate of successful eye drop instillation in the group of subjects who receive the educational session compared to the baseline group subjects (subjects only tested on postoperative day 30 rather than both the first day after surgery and postoperative day 30) who will not receive it.

In comparing the postoperative day 30 proficiency levels of baseline subjects and subjects who were able to proficiently instill a single eye drop on postoperative day 1, the subjects who were able to proficiently instill a single eye drop on postoperative day 1 will have a higher success rate than the baseline group.

The number of subjects who are unable to correctly instill the medication on postoperative day 30 and experienced pain or irritation before or during postoperative day 30 will be higher than the number of subjects who are able to correctly instill the medication on postoperative day 30 and experienced pain or irritation before or during postoperative day 30.

DETAILED DESCRIPTION:
Purpose:

To determine the number of subjects who can proficiently administer one drop of Dexatrol (the steroidal anti-inflammatory drug that Crystal Eye Clinic staff provide to all patients who undergo cataract surgery) on their first attempt on postoperative day 1 and compare this to the number of subjects who can proficiently administer one drop of Dexatrol into the eye that received cataract surgery after using the medication for 30 days.

Baseline/control subjects who are only tested on postoperative day 30 will be referred to as "Group A" subjects. Subjects who will be tested on postoperative day 1 and 30 will be referred to as "Group B" subjects. If "Group B" subjects can proficiently administer the medication on postoperative day 1, they will remain in "Group B" and researchers will determine their rate of success again on postoperative day 30. If subjects cannot proficiently administer the medication on postoperative day 1, they will be re-classified as "Group C" subjects and researchers will determine whether an educational session regarding the correct instillation of eye drops will improve the proficiency of these subjects when they are tested again on postoperative day 30. This will allow staff at Crystal Eye Clinic to understand the effectiveness of their current educational session and will determine the efficacy of an additional educational session. Researchers will also use questionnaires to determine if there are factors that affect the ability of subjects to properly instill the medication as well as if the proficiency of instillation correlates to whether patients experienced irritation or pain before or on postoperative day 30. Dexatrol will not be used outside of its approved indication.

ELIGIBILITY:
Inclusion Criteria:

* Patients who receive cataract surgery sponsored by Unite For Sight from Crystal Eye Clinic from August 20, 2010 to October 2010.
* Patients who had surgery prior to August 20 and will have their postoperative 30 day check up between August 20 and October 20 will be eligible to be Group A subjects.
* Participants must be over 19 and capable of understanding the purpose of the study, risks/benefits involved and all other information needed to provide informed consent.
* Participants must be able to follow instructions (those outlined in the proposal i.e. apply one drop of eye solution into the eye that was operated on).
* Participants must be able to answer the questionnaire either verbally or through writing (with or without the aid of an interpreter).

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People in Ghana needing proficiency of eye drop instillation in postoperative cataract surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Instillation of one drop of Dexatrol into the eye | 30 days
  The primary end-point is the proficiency of patients in instilling one drop of Dexatrol into the eye that received surgery. This will be measured at postoperative day 1 and postoperative day 30 for Group B and C subjects and only postoperative day 30 for Group A subjects.

SECONDARY OUTCOMES:
Irritation or pain after surgery | 30 days
  The secondary end-point is whether subjects feel irritation or pain after surgery. This will be measured on postoperative day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Shafik Dharamsi, Ph.D, Principal Investigator — University of British Columbia; Annalee Yassi, Dr., Study Director — University of British Columbia; Jerry Spiegel, Dr., Study Director — University of British Columbia; Ken Bassett, Dr., Study Director — University of British Columbia; Yang Liu, Dr., Study Director — University of British Columbia; Christian Peoples, Dr., Study Director — University of British Columbia; Tiffany Shiau, Dr., Study Director — University of British Columbia
Locations (1):
- Crystal Eye Clinic, Adenta Housing, No. 5 Giner Close, Accra-North, Ghana